CLINICAL TRIAL: NCT00033150
Title: A Comparison of Language Intervention Programs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U01DC004560 (NIH)
Record Dates: First submitted 2002-04-08; First posted 2002-04-09 (Estimated); Last update posted 2006-04-24 (Estimated); Status verified 2006-04

CONDITIONS: Language Disorders
Keywords: Specific Language Impairment; Fast ForWord; Language therapy; Auditory processing
MeSH Terms: conditions — Language Disorders; Specific Language Disorder

INTERVENTIONS:
Behavioral: Fast ForWord
Behavioral: Computer Assisted Language Intervention
Behavioral: Individual Language Intervention
Behavioral: Academic enrichment

SUMMARY:
Brief Summary:

Nearly 7% of elementary school children present with difficulties learning and using language. Unfortunately, language impairments are often long lasting and may have serious social, academic, and vocational ramifications. More than 1 million children receive language intervention in the public schools each year, and many more are seen in hospitals and other clinical settings.

This randomized clinical trial compares the language outcomes of Fast ForWord to two other interventions (computer assisted language intervention without acoustically modified speech and individual language intervention) and to the outcomes of an academic enrichment (control) condition. Each year for 3 years, children will be randomly assigned to each of the four conditions at three regional sites (Austin, Texas, Dallas, Texas, and Lawrence, Kansas). The treatments will be administered in special summer programs. The primary research question is which intervention results in the most improvement in the composite language score from the Oral and Written Language Scales. Secondary questions include which intervention results in the greatest gains in conversational language,which intervention results in the greatest gains 3 and 6 months after training, which intervention results in the greatest improvement in auditory perception, and which intervention is the most cost effective.

The results of the study will have theoretical and practical value. Theoretically, the study tests the temporal processing hypothesis of language impairment. Practically, the study will describe and compare the language, communication, auditory processing and academic outcomes of different language interventions. The study will help clinicians and administrators choose the most effective and least expensive treatment for the children they serve.

ELIGIBILITY:
Inclusion Criteria:

* age 6 to 9 years
* score between 75 and 125 on the Matrices subtest of the Kaufman Brief Intelligence Test
* Speaking Quotient of 79 or lower on the Test of Language Development: Primary: 3rd Edition

Exclusion Criteria:

* Previous participation in 8 or more hours of language intervention or classroom activities using any of the Fast ForWord, Laureate, or Earobics speech-language or reading software and/or the Lindamood-Bell auditory discrimination training
* Failure of a hearing screening test
* An episode of otitis media in the previous 12 months
* Evidence of focal brain lesion, traumatic brain injury, cerebral palsy, or seizure disorder
* Abnormality of oral structure or function impeding normal language production

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 216
Dates: Start 2002-06; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Gillam, PhD, Principal Investigator — Pflugerville Independent School District
Locations (2):
- United States (2):
  - Lawrence Public Schools USD 497, Lawrence, Kansas
  - Pflugerville Independent School District, Pflugerville, Texas